CLINICAL TRIAL: NCT06275061
Title: Chinese Obesity and MEtabolic Surgery Database
Brief Title: Chinese Obesity and MEtabolic Surgery Database (COMES Database)
Acronym: COMES
Status: Recruiting | Type: Observational
Sponsor: Jinan University Guangzhou (Other)
Collaborators: Chinese Obesity and Metabolic Surgery Collaborative (Unknown)
Responsible Party: Principal Investigator, Wah Yang, MD, Principal Investigator, Jinan University Guangzhou
Other Study IDs: KY-2020-021
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Metabolic Surgery; Bariatric Surgery; Weight Loss
Keywords: Obesity; Metabolic Surgery; Bariatric Surgery; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Metabolic Networks and Pathways; Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metabolic and Bariatric Surgery: Metabolic and bariatric surgery is weight loss surgery that results in weight loss and resolution of metabolic disorders.
  Interventions: Procedure: Metabolic and Bariatric Surgery

INTERVENTIONS:
Procedure: Metabolic and Bariatric Surgery — Metabolic and bariatric surgery is weight loss surgery that results in weight loss and resolution of metabolic disorders.

SUMMARY:
The purpose of the Chinese Obesity and MEtabolic Surgery Database (COMES Database) is to collect data and examine the long-term effects of metabolic and bariatric surgery on obesity and metabolic disorders in the Chinese population.

DETAILED DESCRIPTION:
COMES Database is a prospective managed national database to collect data and examine the long-term effects of metabolic and bariatric surgery on obesity and metabolic disorders in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as obesity undergoing metabolic and bariatric surgery.

Exclusion Criteria:

* Patients treated by non-surgical modalities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed as obesity undergoing metabolic and bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Excess weight loss effect of metabolic and bariatric surgery after 1 year | 1 year
  Percent excess weight loss (%EWL) = [(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)]

SECONDARY OUTCOMES:
Excess weight loss effect of metabolic and bariatric surgery in long-term follow-ups | 3 years
  Percent excess weight loss (%EWL) = [(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)]
Excess weight loss effect of metabolic and bariatric surgery in long-term follow-ups | 5 years
  Percent excess weight loss (%EWL) = [(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)]
Excess weight loss effect of metabolic and bariatric surgery in long-term follow-ups | 10 years
  Percent excess weight loss (%EWL) = [(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)]
Glycemic control effect of metabolic and bariatric surgery after 1 year | 1 year
  Change of HbA1c levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 3 years
  Change of HbA1c levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 5 years
  Change of HbA1c levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 10 years
  Change of HbA1c levels
Glycemic control effect of metabolic and bariatric surgery after 1 year | 1 year
  Change of blood glucose levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 3 years
  Change of blood glucose levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 5 years
  Change of blood glucose levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 10 years
  Change of blood glucose levels
Glycemic control effect of metabolic and bariatric surgery after 1 year | 1 year
  Change of C-peptide levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 3 years
  Change of C-peptide levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 5 years
  Change of C-peptide levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 10 years
  Change of C-peptide levels
Glycemic control effect of metabolic and bariatric surgery after 1 year | 1 year
  Change of insulin levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 3 years
  Change of insulin levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 5 years
  Change of insulin levels
Glycemic control effect of metabolic and bariatric surgery in long-term follow-ups | 10 years
  Change of insulin levels

OTHER OUTCOMES:
Adverse events rate of metabolic and bariatric surgery | 30 days after surgery
  Surgical safety by 30 days follow-up according to guideline

CONTACTS AND LOCATIONS:
Overall Officials: Cunchuan Wang, MD, PhD, Study Chair — First Affiliated Hospital of Jinan University; Wah Yang, MD, Study Director — First Affiliated Hospital of Jinan University
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No